CLINICAL TRIAL: NCT05438381
Title: Assistant Lecturer of Pediatric Dentistry, Mansoura University (2019)
Brief Title: Comparison of Clinical and Radiographic Outcomes of SMART Technique vs ART in Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A 04030919
Record Dates: First submitted 2022-05-10; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Dental Caries
Keywords: SDF; ART; SMART technique
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ART group (Active Comparator): Atraumatic restorative technique: excavation of caries then application of Glass ionomer capsule (GC, USA)
  Interventions: Procedure: Atraumatic Restorative Technique (ART)
- SMART group (Experimental): SMART technique: excavation of caries and application of silver diamine fluoride (SDF 38%) then glass ionomer cement
  Interventions: Procedure: SMART Technique

INTERVENTIONS:
Procedure: Atraumatic Restorative Technique (ART) — Glass ionomer capsule (GC, USA)
  Arms: ART group
Procedure: SMART Technique — silver diamine fluoride (SDF) then glass ionomer cement capsule (GC, USA)
  Arms: SMART group

SUMMARY:
This study conducted on thirty children aged 3-6 years old of both genders, have bilateral carious lower first primary molars. Pre-operative periapical x- ray were taken for both sides. The children were divided into 2 groups(SMART group and ART group). For Atraumatic Restorative Technique (ART technique), glass ionomer cement(GIC) was applied according to manufacturer's instructions. For Silver Modified Atraumatic Restorative Technique (SMART technique), SDF was applied carefully using bended micro sponge brush. It was applied directly to only the affected tooth surface. After one week GIC was applied according to manufacturer's instructions. Clinical and radiographic evaluation were done for all teeth at 6, 12 months. The data were collected then statistically analyzed using chi-square test to show the difference between groups.

DETAILED DESCRIPTION:
Sample size calculation:

For this study, a sample size of 30 was obtained using unpaired two sample two tail z-test. The effect size (dz=2.813) and the required sample size were calculated for α =0.05 and a confidence power of 0.8039, assuming a normal distribution.

Patient selection: This study conducted on thirty children aged 3-6 years old of both genders. The children selected from Pediatric Dental Clinic, Faculty of Dentistry, Mansoura University. Included children in the study were. Apparent healthy and free from any systemic diseases or chronic conditions. Child should have bilateral restorable carious lower first primary molars, occlusal caries, International Caries Detection and Assessment System(ICDAS) score (4, 5), asymptomatic or have reversible pulpitis. Radiographic examination show intact lamina dura, absence of internal and external pathological root resorption or periapical infection.

Randomization. The study was spilt mouth design. The right side of all participants was done atraumatic restorative technique (ART) and the left side was silver modified atraumatic restorative technique (SMART technique).

Clinical procedures:

* Communication with the children were established.
* Pre-operative periapical x- ray were taken for both sides.
* Gross debris from cavitation were removed.
* Carious dentin on walls were excavated using spoon excavator and low speed contra with round or fissure bur.
* Areas to be treated were isolated with cotton rolls.
* Dryness of lesion with gentle flow of compressed air were done. Control group: Right side of the patient (ART technique) (group 1) (D1) :(20)
* GIC was applied according to manufacturer's instructions.

Experimental group: Left side of the patient (SMART technique) (group 2) (D2):(21)

* A protective coating was applied to the lips and skin to prevent a temporary henna-appearing tattoo that can occur if soft tissues come into contact with SDF.
* SDF was applied carefully using bended micro sponge brush. The brush was dipped into SDF and dabbed on the side of the plastic dish to remove excess liquid before application.
* SDF was applied directly to only the affected tooth surface of lower first primary molar.
* Excess SDF was removed with gauze, cotton roll, or cotton pellet to minimize systemic absorption.
* Application time was at least one minute. No more than one drop of SDF was used for the entire appointment.
* The lesion was dried for 15 seconds with gentle flow of compressed air.
* After one week GIC was applied according to manufacturer's instructions.

Evaluation:

All primary molars were evaluated clinically and radiographically at 6 and 12 months for the overall success/failure criteria:

* Presence/absence of {recurrent caries (catch with probe), pain (spontaneous, with eating, with percussion), clinical abscess, mobility}.
* Presence/absence of {internal root resorption, external root resorption, interradicular radiolucency, periapical radiolucency}.

Statistical Analysis:

The collected data were tabulated and statistically analyzed . The results were considered statistically significant at p≤0.05.

* Chi-Square test was performed to compare the significance between the groups in clinical and radiographic evaluation.
* Kappa index was performed to correlate between clinical and radiographic results.

ELIGIBILITY:
Inclusion Criteria:

* This study conducted on thirty children aged 3-6 years old of both genders.
* children in the study were. Apparent healthy and free from any systemic diseases or chronic conditions.
* Child should have bilateral restorable carious lower first primary molars, occlusal caries, ICDAS score (4, 5), asymptomatic or have reversible pulpitis.
* Radiographic examination show intact lamina dura, absence of internal and external pathological root resorption or periapical infection.

Exclusion Criteria:

-

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
post operative pain | 12 months
  numerical/visual analogue scale 0 no pain 10 worst possible pain
radiolucency | 12 months
  x ray will be done( qualitative assessment looking for presence of interradicular or periapical radiolucency will be performed and will be scored as yes or no)
Pathological internal or external root resorption | 12 months
  x ray will be done( qualitative assessment looking for presence of pathological internal or external root resorption will be performed and will be scored as yes or no)

SECONDARY OUTCOMES:
tooth mobility | 12 months
  clinical method of assessing tooth mobility 0 no mobility 3 mobility more than 2 mm bucco-lingually
Presence or absence of fistula | 12 months
  visual inspection( visual assessment will be performed clinically looking for presence or absence and will be scored yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: sahar mohammed, dentist, Principal Investigator — Mansoura University
Locations (1):
- University, Al Mansurah, El Gomhoria Street, Mansoura,egypt, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Contreras V, Toro MJ, Elias-Boneta AR, Encarnacion-Burgos A. Effectiveness of silver diamine fluoride in caries prevention and arrest: a systematic literature review. Gen Dent. 2017 May-Jun;65(3):22-29. PMID 28475081